CLINICAL TRIAL: NCT04367272
Title: Is Second Knee at Risk During Simultaneous Bilateral Total Knee Arthroplasty.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, Residents Doctor in Orthopedics Department, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27.04.2020-02
Record Dates: First submitted 2020-04-25; First posted 2020-04-29 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis, Knee; Infection; Periprosthetic Fracture Around Prosthetic Joint Implant
MeSH Terms: conditions — Osteoarthritis, Knee; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Knee (Active Comparator): The first knee is the knee where the surgery will begin to be applied.
  Interventions: Procedure: First Arthroplasty
- Second Knee (Experimental): The second knee is the knee where the surgeon will apply secondly.
  Interventions: Procedure: Second Arthroplasty

INTERVENTIONS:
Procedure: First Arthroplasty — First Knee
  Arms: First Knee
Procedure: Second Arthroplasty — Second Knee
  Arms: Second Knee

SUMMARY:
The effects of single-team simultaneous bilateral total knee arthroplasty on peri- and postoperative complications are clear. The investigators hypothesized that second knee at risk during single-team simultaneous bilateral total knee arthroplasty and have more early postoperative complication rates than the first knee. Therefore, this prospective study compared minor and major local complications for 90 days postoperatively between the first and second during knee single-team simultaneous bilateral total knee arthroplasty.

DETAILED DESCRIPTION:
The investigators would like to compare operation related technical complications and periprosthetic joint infection rate between the first and second knee.

ELIGIBILITY:
Inclusion Criteria:

* Primary bilateral knee osteoarthritis with refractory to conservative treatment
* Patients who accept participation in the research and the randomization

Exclusion Criteria:

* no history of malignancy
* less than 75 years old
* severe cardiac insufficiency and morbid obesity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Local complications | 90 days
  Local operation related complications rate

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR